CLINICAL TRIAL: NCT05612763
Title: Self Fitting Hearing Aid Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Starkey Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GQ-PRO-06093
Record Dates: First submitted 2022-10-28; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Hearing Loss, Sensorineural
Keywords: self fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: The participants will have three lab sessions and two field trials. In the first session, every participant will receive PD and CD fittings. The wearing schedule orders for all the participants will be counterbalanced. For the first field trial, half of the participants will wear the hearing aids with PD and the other half of the participants will wear the hearing aids with CD. In session two, outcomes for the first hearing aid condition will be measured. Then, the participants will wear hearing aids with the other type of fitting strategy for the second field trial. After that, they will return to the lab for session 3, in which outcomes for the second hearing aid condition will be measured. Outcome measures include a self-report field evaluation (Abbreviated Profile of Hearing Aid Benefit, or APHAB) and a lab-based speech recognition test (Quick Speech-in-Noise Test, Quick-SIN).
Masking Description: participant is not told which fitting method they have been assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Method of fit (Experimental): Devices are fit using either a clinician completed fitting process or a patient completed fitting process. Then the alternate fitting method is used to repeat the process. The order of which method used is counterbalanced.
  Interventions: Device: Self fitting hearing device

INTERVENTIONS:
Device: Self fitting hearing device — comparison of outcomes when device is fit by clinician or self fit

SUMMARY:
Pre-market Clinical Investigation whose primary purpose is to evaluate efficacy and effectiveness of self-fitting hearing aids

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the outcomes of hearing aids with patient-driven fitting (PD) and clinician-driven fitting (CD). The participants will be 40 adults with mild to moderate symmetrical hearing loss. For each hearing aid fitting strategy, the participant will wear the hearing aids for 10 days. Lab and field outcomes will be measured. This study will determine if perceived hearing benefit and speech recognition performance with the PD fitting method is non-inferior to that with the CD fitting method.

ELIGIBILITY:
Inclusion Criteria:

1. Native English speakers
2. Ability to complete questionnaires and laboratory assessments
3. Symmetric, mild to moderate sensorineural hearing loss
4. Informed consent completed with signature
5. Healthy outer ear/middle ear status
6. Limited hearing aid use (non-owners of hearing aids)

Exclusion criteria:

1. Inability to visit the Starkey Headquarters building for testing
2. Central or middle ear hearing pathology
3. Medical contraindications to wearing hearing aids
4. Learning disability, major cognitive handicap, or serious neurological or psychiatric disease that would prevent or restrict participation, as determined by the PI or designee
5. Hearing loss outside of the specified criteria (Mild to Moderate Sensorineural hearing loss)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
1. Perceived hearing aid benefit- Abbreviated Profile of Hearing Aid Benefit (APHAB) | The timeframe for this data collection will be unaided, and 14 days post-fitting.
  This data will be collected through the APHAB (Abbreviated Profile of Hearing Aid Benefit). This is a 24-item survey of hearing aid benefit. This test will be administered in the unaided hearing aid condition, and in both the traditional and new fitting method conditions. Scores report the reduction in reported problems, and a higher score shows a larger reduction in problems in one condition than the other.

SECONDARY OUTCOMES:
1. Speech intelligibility - Quick Speech in Noise Test (QuickSIN) | Timeframe for this data collection will be unaided, and 14-days post-fitting.
  This data will be collected with the QuickSIN, which is an adaptive measure of speech recognition in background noise. Outcome score is reported in "dB SNR loss." A reduced SNR loss is a better score and implies that the lower score performs better than the higher score.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hicks, PhD, Study Director — VP education and Clinical Studies
Locations (1):
- Starkey Laboratories, Eden Prairie, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Overall data that does not identify the individual will be made available upon request, and summaries of the study data and data analysis will be provided